CLINICAL TRIAL: NCT03492047
Title: Evaluation of The Effect of N-AcetylCysteine in The Prevention of Paclitaxel-Induced Peripheral Neuropathy in Cancer Patients
Brief Title: N-acetyl Cysteine Effect in Peripheral Neuropathy in Cancer Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Nasser Institute For Research and Treatment (Other Government)
Responsible Party: Principal Investigator, Hadeer Gamal Khalefa, pharmacist, Nasser Institute For Research and Treatment
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHCL93
Record Dates: First submitted 2018-03-02; First posted 2018-04-10 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Peripheral Neuropathy Due to Chemotherapy
Keywords: paclitaxel; peripheral neuropathy; N-acetyl cysteine
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Acetylcysteine; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Active Comparator): they will receive paclitaxel 80 mg/m2 once per week for 12 weeks only
  Interventions: Drug: Paclitaxel
- high dose N-acetyl cysteine (Experimental): they will receive paclitaxel 80 mg/m2 once per week for 12 weeks and high dose N-acetylcysteine (1200 mg twice daily) for the paclitaxel treatment period
  Interventions: Dietary Supplement: high dose N-acetylcysteine; Drug: Paclitaxel
- low dose N-acetyl cysteine (Experimental): they will receive paclitaxel 80 mg/m2 once per week for 12 weeks and low dose N-acetylcysteine (600mg twice daily) for the paclitaxel treatment period.
  Interventions: Dietary Supplement: low dose N-acetylcysteine; Drug: Paclitaxel

INTERVENTIONS:
Dietary Supplement: low dose N-acetylcysteine — N-acetylcysteine 600mg twice daily
  Arms: low dose N-acetyl cysteine
Dietary Supplement: high dose N-acetylcysteine — N-acetylcysteine 1200mg twice daily
  Arms: high dose N-acetyl cysteine
Drug: Paclitaxel — Paclitaxel 80mg /m2 IV

SUMMARY:
The purpose of the study is to evaluate the effect of N-acetyl cysteine in combination with paclitaxel on the clinical outcomes of patients with peripheral neuropathy, paclitaxel-induced peripheral neuropathy affect quality of life in cancer patients.

new therapeutic approches such as the antioxidant N-acetyl cysteine, showed to has neuroprotective effect, the aim of the study is to evaluate the effect of N- acetylcysteine(NAC) administration in the prevention of paclitaxel-Induced peripheral neuropathy.

DETAILED DESCRIPTION:
Paclitaxel is a first-line chemotherapeutic treatment of solid tumors. Neuronal damage also seems to have a major role in paclitaxel-induced neuropathic pain, paclitaxel contributes to ROS formation (superoxide, hydroxyl radical, nitric oxide and hydrogen peroxide) in neuronal mitochondria that are involved in nerve injury-induced.

N-acetylcysteine (NAC) is a cysteine pro-drug and glutathione (GSH) precursor which is a protective agent and detoxifies and scavenges reactive oxygen species (ROS), which seems to help normalize the oxidative status.

It has been reported that high dose of N-acetylcysteine shown to Prevent retrograde motor neuron death after neonatal peripheral nerve injury and significantly increases motor neuron survival, which may improve functional outcomes after obstetrical brachial plexus injury in rats.

Also, it has been reported that NAC significantly inhibited CCI-induced microglia activation but elicited no notable effects on astrocytes. These results demonstrate an effective and safe approach that has been used clinically to alleviate neuropathic pain via the powerful inhibition of the activation of MMPs in rats.

N-acetylcysteine has been shown to have neuroprotective effects against oxaliplatin-based adjuvant chemotherapy in colon cancer patients with Oral administration of N-acetylcysteine1,200 mg) was given one and a half hours before each oxaliplatin administration.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>18 years old).
2. Breast cancer patients who will receive adjuvant weekly paclitaxel for 12 cycles.
3. ECOG performance status 0-2
4. Adequate bone marrow function (white blood count ≥4,000/mm3, platelet count ≥100,000/mm3), liver function (serum total bilirubin <1.5 mg/dl), renal function (creatinine <1.5 mg/dl).

Exclusion Criteria:

1. Patients who have any of the following:

   * Clinical neuropathy.
   * Diabetes mellitus.
2. Patients receiving vitamin B1, B6, B12,or other vitamin supplemental therapy.
3. Patients receiving antidepressants, opioids, adjuvant analgesic agents (eg, anticonvulsants, clonazepam, or mexiletine), topical analgesics, and amifostine.
4. Hypersensitivity to NAC.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence of chemotherapy induced-peripheral neuropathy | up to 12 week
  Number of patients reported neuropathy from paclitaxel

SECONDARY OUTCOMES:
severity of chemotherapy induced-peripheral neuropathy | at baseline and before each cycle up to 12 week
  severity of paclitaxel induced peripheral neuropathy using NCI-CTCAE criteria
Adverse effects | at baseline and each cycle up to 12 week
  any adverse/ side effect will be evaluated
severity of chemotherapy induced-peripheral neuropathy | at baseline, at the end of 6 cycle and at the end of 12 cycles
  severity of chemotherapy induced-peripheral neuropathy using modified total neuropathy score ,Each neuropathy item is scored by a physician on a 0-4 scale the scores are summed to obtain a total score, modified total neuropathy score score ranges from 0-24 with higher total scores indicate more severe neuropathy.

OTHER OUTCOMES:
the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group-Neurotoxicity(FACT-GOG-NTX) subscale | weekly up to 12 week
  measures quality of life related to signs and symptoms of paclitaxel induced peripheral neuropathy
serum nerve growth factor | at baseline and after 12 week
  measuring serum level of nerve growth factor using ELISA KIT
serum malionaldehyde | at baseline and after 12 week
  measuring serum level of maliomaldehyde using spectrophometric kit

CONTACTS AND LOCATIONS:
Overall Officials: Hadeer G Khalefa, master, Principal Investigator — Nassar institute for research and treatment hospital
Locations (1):
- AinShams University Hospitals, Cairo, Egypt

REFERENCES:
- [Derived] Khalefa HG, Shawki MA, Aboelhassan R, El Wakeel LM. Evaluation of the effect of N-acetylcysteine on the prevention and amelioration of paclitaxel-induced peripheral neuropathy in breast cancer patients: a randomized controlled study. Breast Cancer Res Treat. 2020 Aug;183(1):117-125. doi: 10.1007/s10549-020-05762-8. Epub 2020 Jun 29. PMID 32601973